CLINICAL TRIAL: NCT03635879
Title: A Phase 1, Single-Center, Pilot, Single-Dose, 6-Way Crossover Study to Compare Six Formulations of Medium Chain Triglycerides on the Pharmacokinetics of Ketone Body Production
Brief Title: Medical Food Formulation Pharmacokinetic (PK) Study in Medium Chain Triglycerides
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study redesign
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AX-18-018_PK
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — AC-1202

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- MCTprocal medical food (Active Comparator): Vitaflo MCTprocal, single dose (20 g MCT)
  Interventions: Other: MCTprocal medical food
- Milk/tricaprilin oil blend (Active Comparator): Lactose-free milk and tricaprilin oil, blended,single dose (20 g tricaprilin)
  Interventions: Other: Milk/tricaprilin oil blend
- AC-1207 (Active Comparator): AC-1207 liquid, single dose (20 g tricaprilin)
  Interventions: Other: AC-1207
- AC-1205 (Active Comparator): AC-1205 liquid, single dose (20 g tricaprilin)
  Interventions: Other: AC-1205
- AC-1206 (Active Comparator): AC-1206 liquid, single dose (20 g tricaprilin)
  Interventions: Other: AC-1206
- AC-1202 (Experimental): AC-1206 liquid, single dose (20 g tricaprilin)
  Interventions: Drug: AC-1202

INTERVENTIONS:
Other: MCTprocal medical food — 32 g MCTprocal (20 g MCT) mixed in 180 mL of water at Hour 0 Day 1
  Arms: MCTprocal medical food
Other: Milk/tricaprilin oil blend — 154 mL of lactose-free skim milk/21 mL of tricaprilin oil blended and then mixed in 180 mL of water at Hour 0 Day 1
  Arms: Milk/tricaprilin oil blend
Other: AC-1207 — AC-1207 (20 g MCT) mixed in 180 mL of water at Hour 0 Day 1
  Arms: AC-1207
Other: AC-1205 — AC-1205 (20 g MCT) mixed in 180 mL of water at Hour 0 Day 1
  Arms: AC-1205
Other: AC-1206 — AC-1206 (20 g MCT) mixed in 180 mL of water at Hour 0 Day 1
  Arms: AC-1206
Drug: AC-1202 — AC-1202 (20 g MCT) mixed in 240 mL of water at Hour 0 Day 1
  Arms: AC-1202

SUMMARY:
This is a Phase I, open label, randomized, 6-way crossover, pilot PK study

DETAILED DESCRIPTION:
12 healthy, male subjects enrolled, subject will be randomized to receive a single dose of one of six treatment, with a 2 day washout in between each dosing period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male 18 55 years of age, inclusive, at Screening.
2. Continuous non smoker who has not used nicotine containing products for at least 3 months prior to Day -1 of Period 1 and throughout the study based on self-reporting.
3. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at Screening.
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee. At screening, subjects must have alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) ≤ the upper limit of normal and triglyceride levels must be < 250 mg/dL.
5. Hemoglobin levels ≥ the lower limit of normal at Screening and Day -1 of Period 1.
6. A non vasectomized subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to Day -1 of Period 1. A subject who has been vasectomized less than 4 months prior to Day -1 of Period 1 must follow the same restrictions as a non vasectomized male).
7. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past year prior to Day -1 of Period 1.
5. History or presence of galactosemia or hypersensitivity or idiosyncratic reaction to the study drugs, related compounds, milk, palm or coconut oil, or soy.
6. History or presence of symptomatic diverticular disease, uncontrolled gastroesophageal reflux disease, ulcers, inflammatory bowel disease, irritable bowel syndrome or recurrent diarrhea, or gout.
7. Positive urine drug results at Screening or Check-in.
8. Positive alcohol results at Screening or Check-in. One repeat assessment is permitted.
9. Positive results at Screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
10. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at Screening. One repeat assessment is permitted.
11. Seated heart rate is lower than 40 bpm or higher than 99 bpm at Screening.
12. QTcF interval is >460 msec or subject has ECG findings deemed abnormal with clinical significance by the PI or designee at Screening.
13. Estimated creatinine clearance ≤ 80 mL/min at Screening.
14. Unable to refrain from or anticipates the use of any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to Day -1 of Period 1 and throughout the study. Acetaminophen (up to 2 g per 24 hours) may be permitted during the study.
15. Has been on a diet incompatible with the on-study diet, in the opinion of the PI or designee, within the 28 days prior to Day -1 of Period 1 and throughout the study.
16. Has been following a ketogenic diet, in the opinion of the PI or designee, within 2 weeks prior to Day -1 of Period 1.
17. Is lactose intolerant.
18. Is unable to complete the standard breakfast prior to dosing on Day 1 of each Period.
19. Donation of blood or significant blood loss within 56 days prior to Day -1 of Period 1.
20. Plasma donation within 7 days prior to Day -1 of Period 1.
21. Participation in another clinical study within 28 days prior to Day -1 of Period 1. The 28-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day -1 of Period 1 of the current study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-13 (Estimated); Primary Completion 2019-04-16 (Estimated); Study Completion 2019-04-16 (Estimated)

PRIMARY OUTCOMES:
Total ketones | 1 day
  Area Under the Curve (AUC) AUC 0 - last
Total ketones | 1 day
  AUC 0 - 4
Total ketones | 1 day
  AUC 0 - 6
Total ketones | 1 day
  AUC 0 - 8
Total ketones | 1 day
  Maximum Plasma Concentration (Cmax)
B-hydroxybutyrate | 1 day
  AUC 0 - last
B-hydroxybutyrate | 1 day
  AUC 0 - 4
B-hydroxybutyrate | 1 day
  AUC 0 - 6
B-hydroxybutyrate | 1 day
  AUC 0 - 8
B-hydroxybutyrate | 1 day
  Cmax
Acetoacetate | 1 day
  AUC 0 - last
Acetoacetate | 1 day
  AUC 0 - 4
Acetoacetate | 1 day
  AUC 0 - 6
Acetoacetate | 1 day
  AUC 0 - 8
Acetoacetate | 1 day
  Cmax

IPD SHARING:
Plan to Share IPD: No